CLINICAL TRIAL: NCT06653530
Title: Efficacy and Safety of Thread Embedding Acupuncture Therapy for Weight Loss in Adults with Overweight or Obesity
Brief Title: Thread Embedding Acupuncture Therapy for Weight Loss
Acronym: iSho
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Li bin, Professor, Beijing Hospital of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024BL02-055-02
Record Dates: First submitted 2024-10-21; First posted 2024-10-22 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2024-10

CONDITIONS: Obesity and Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Thread embedding acupuncture (Experimental): The participants in the thread embedding acupuncture therapy group will receive treatment that consists of 18 thread embedding acupuncture sessions over a 24-week period after baseline (once a week for the first 12 weeks and every two weeks for the next 12 weeks).
  Interventions: Other: Thread embedding acupuncture
- Sham thread embedding acupuncture (Sham Comparator): The participants in the sham thread embedding acupuncture therapy group will receive treatment that consists of 18 sham thread embedding acupuncture sessions over a 24-week period after baseline (once a week for the first 12 weeks and every two weeks for the next 12 weeks).
  Interventions: Other: Sham thread embedding acupuncture

INTERVENTIONS:
Other: Thread embedding acupuncture — Thread embedding acupuncture is performed using polyglycolic acido thread. Needles have a gauge size of 23G, a shaft length of 60mm, and a thread length of 50mm, folded in half, and are applied to fourteen acupoints, including Zhongwan (CV12), Qihai (CV6), bilateral Tianshu (ST 25), bilateral Wailing (ST 26), bilateral Daheng (SP 15), bilateral Zusanli (ST 36), bilateral Pishu (BL 20), and bilateral Weishu (BL 21). After the thread is inserted into the body, the needle will be withdrawn immediately. During the treatment period, health counseling will be provided by qualified staff at every visit, including diet and physical activity, but there will be no strict restrictions.
  Arms: Thread embedding acupuncture
Other: Sham thread embedding acupuncture — The protocol includes the same duration and frequency of sessions as for thread embedding acupuncture, but the treatment will be delivered superficially at non-acupuncture points 10mm from the lateral of the corresponding acupuncture and not above a meridian line. Needles without threads have a gauge size of 23G, and a shaft length of 60mm will be used. After the needle is inserted into the body, it will be withdrawn immediately. During the treatment period, health counseling will be provided by qualified staff at every visit, including diet and physical activity, but there will be no strict restrictions.
  Arms: Sham thread embedding acupuncture

SUMMARY:
Obesity is the most prevalent chronic disease worldwide, affecting approximately 800 million adults. Excess adiposity and its numerous complications, including cardiovascular disease and type 2 diabetes, impose a considerable economic burden and constitute major contributors to global morbidity and mortality. Treatments that result in substantial weight reductions may improve outcomes for people living with obesity. Thread embedding acupuncture which provides long-term acupoints stimulation may be an effective treatment option for obesity. However, effects of thread embedding on obesity remain uncertain because of the small sample sizes or other methodological limitations. The objective of this multi-center, randomized, sham-controlled trial is to assess the effect of thread embedding acupuncture for alleviating weight.

DETAILED DESCRIPTION:
The present multi-center, randomized, sham-controlled, parallel-group trial aims to evaluate the effect of thread embedding acupuncture in patients with obesity.

The patients will be randomized to receive one of two treatment arms: thread embedding acupuncture and sham thread embedding acupuncture. The participants will receive treatment that consists of 18 thread embedding acupuncture or sham thread embedding acupuncture sessions over a 24-week period after baseline (once a week for the first 12 weeks and every two weeks for the next 12 weeks). At the end of 24 weeks treatment, the change of weight in overweight/obese participants between the two groups will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Body-mass index: a. BMI ≥ 28 kg/m2 or b. BMI ≥ 24 kg/m2 with the presence of at least one of the following weight-related complications (treated or untreated): diabetes, hypertension, lipid metabolism disorders, obstructive sleep apnea, cardiovascular disease, knee osteoarthritis, hyperuricemia, fatty liver;
2. Male or female, age between 18 and 75 years at the time of signing informed consent;
3. No history of receiving thread embedding treatment;
4. History of at least one self-reported unsuccessful dietary effort and exercise program to lose body weight;
5. Informed consent obtained.

Exclusion Criteria:

1. A self-reported change in body weight ≥ 5 kg within 90 days before screening;
2. Treatment with any medication for the indication of obesity within the past 90 days before Screening;
3. Previous or planned (during the trial period) obesity treatment with surgery or a bodyweight loss device. However, the following were allowed: (1) liposuction and/or abdominoplasty, if performed more than 1 year before screening; (2) lap banding, if the band had been removed more than 1 year before screening; (3) intragastric balloon, if the balloon had been removed more than 1 year before screening; or (4) duodenal-jejunal bypass sleeve, if the sleeve had been removed more than 1 year before screening;
4. Have obesity induced by other endocrinologic disorders (for example, Cushing Syndrome) or diagnosed monogenetic or syndromic forms of obesity (for example, Melanocortin 4 Receptor deficiency or Prader Willi Syndrome);
5. Uncontrolled thyroid disease, defined as thyroid stimulating hormone (TSH)>6.0 mIU/L or <0.35 mIU/L as measured by the central laboratory at screening;
6. Diagnosed with type 2 diabetes mellitus ≤180 days prior to the day of screening or those who have taken treatment with oral agents that were unstable (different drug(s), dose, or dosing frequency) within the 90 days prior to screening;
7. Receipt of any acupuncture treatment for obesity within 90 days before screening;
8. Participation in any structured, monitored weight-loss program within 90 days before screening;
9. Active inflammatory bowel disease, celiac disease, chronic pancreatitis, or other disorder potentially causing malabsorption;
10. Any of the following severe cardiovascular diseases: myocardial infarction, stroke, heart failure, symptomatic peripheral vascular diseases, or hospitalization for unstable angina or transient ischemic attack within the last 6 months prior to screening;
11. History of malignant neoplasms within the past 5 years prior to screening. Basal and squamous cell skin cancer and any carcinoma in-situ are allowed;
12. Chronic respiratory, neurological, musculoskeletal or other disorders where, in the judgement of the investigator, participants would have unacceptable risk or difficulty in complying with the protocol;
13. Surgery scheduled for the duration of the trial, except for minor surgical procedures, in the opinion of the investigator;
14. Known or suspected abuse of alcohol or recreational drugs;
15. Female who was pregnant, breast-feeding, or intended to become pregnant, or was of child-bearing potential and not using a highly effective contraceptive method;
16. Known or suspected hypersensitivity to trial product or related products;
17. Participation in another clinical trial within 90 days before screening;
18. Any disorder, unwillingness, or inability, not covered by any of the other exclusion criteria, which in the investigator's opinion might have jeopardised the participant's safety or compliance with the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Relative change in body weight | From baseline (week 0) to end of treatment (week 24)
  Measured in percentage (%)

SECONDARY OUTCOMES:
Body weight reduction greater than or equal to 5% | From baseline (week 0) to end of treatment (week 24)
  Measured as the percentage of participants
Body weight reduction greater than or equal to 10% | From baseline (week 0) to end of treatment (week 24)
  Measured as the percentage of participants
Change in body weight | From baseline (week 0) to end of treatment (week 24)
  Measured in kilogram (kg)
Change in Body Mass Index (BMI) | From baseline (week 0) to end of treatment (week 24)
  Measured in kilogram per square meter (kg/m^2)
Change in body fat rate | From baseline (week 0) to end of treatment (week 24)
  Measured in percentage points
Change in waist circumference | From baseline (week 0) to end of treatment (week 24)
  Measured in centimeter (cm)
Change in waist-to-hip ratio | From baseline (week 0) to end of treatment (week 24)
  Calculated by dividing the waist circumference(cm) by the hip circumference(cm).
Change in Systolic Blood Pressure (SBP) | From baseline (week 0) to end of treatment (week 24)
  Measured in millimeter of mercury (mmHg)
Change in Diastolic Blood Pressure (DBP) | From baseline (week 0) to end of treatment (week 24)
  Measured in mmHg
Change in Glycated Haemoglobin (HbA1c) | From baseline (week 0) to end of treatment (week 24)
  Measured in percentage points
Change in Fasting Plasma Glucose (FPG) | From baseline (week 0) to end of treatment (week 24)
  Measured as millimole per liter (mmol/L)
Change in fasting serum insulin | From baseline (week 0) to end of treatment (week 24)
  Measured as milli-international units per milliliter (mIU/mL)]
Change in high-density lipoprotein (HDL) cholesterol | From baseline (week 0) to end of treatment (week 24)
  Measured as mmol/L
Change in low-density lipoprotein (LDL) cholesterol | From baseline (week 0) to end of treatment (week 24)
  Measured as mmol/L
Change in triglycerides | From baseline (week 0) to end of treatment (week 24)
  Measured as mmol/L
Change in total cholesterol | From baseline (week 0) to end of treatment (week 24)
  Measured as mmol/L
Change in Short Form-36 (SF- 36) Physical Functioning score | From baseline (week 0) to end of treatment (week 24)
  The SF-36 is a 36-item commonly used generic clinical outcome assessment instrument measuring health-related quality of life and general health status across disease areas. SF-36 questionnaire measures 8 domains of functional health and well-being as well as 2 component summary scores (physical component summary and mental component summary). This endpoint assesses the physical functioning domain.
Change in SF-36: Physical Component Summary Score | From baseline (week 0) to end of treatment (week 24)
  The SF-36 is a 36-item commonly used generic clinical outcome assessment instrument measuring health-related quality of life and general health status across disease areas. SF-36 questionnaire measures 8 domains of functional health and well-being as well as 2 component summary scores (physical component summary and mental component summary).This endpoint assesses the physical component summary.
Change in SF-36: Mental Component Summary score | From baseline (week 0) to end of treatment (week 24)
  The SF-36 is a 36-item commonly used generic clinical outcome assessment instrument measuring health-related quality of life and general health status across disease areas. SF-36 questionnaire measures 8 domains of functional health and well-being as well as 2 component summary scores (physical component summary and mental component summary). This endpoint assesses the mental component summary.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Hospital of Traditional Chinese Medicine, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No